CLINICAL TRIAL: NCT06462716
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of BY101298 as Single-agent Therapy/in Combination With Radiotherapy in Patients With Malignant Solid Tumors
Brief Title: A Phase l Study of By101298, an Oral DNA-PK Inhibitor, in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Baiyu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BY1298-I-01
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BY101298 (Experimental): Dose Escalation: Subjects will receive a starting dose of 50 milligram (mg) of BY1298 as Capsule orally once daily, ascending to 100, 200, 300 and 400 mg. If MTD is not reached at 400 mg, other dosage will be explored.
  Interventions: Drug: BY101298 Capsules

INTERVENTIONS:
Drug: BY101298 Capsules — An oral DNA-PK Inhibitor

SUMMARY:
BY101298 is an innovative DNA-dependent protein kinases (DNA-PK) highly selective small molecule inhibitor. DNA-dependent protein kinases (DNA-PK plays a key role in the NHEJ repair pathway to repair DNA double-strand breaks (DSBs).

Primary objective is to assess the safety and tolerability of BY101298 in patients with advanced malignant solid tumors. The secondary Objectives are to characterize the pharmacokinetic (PK) profile of BY101298 in patients with advanced malignant solid tumors and to assess the preliminary efficacy of BY101298 in patients with advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, ≥ 18 and ≤ 75 years of age (inclusive at the time of informed consent).
2. Diagnostic outcome:

   Phase Ia: patients histologically or cytologically diagnosed advanced malignant solid tumors who have failed, cannot tolerate, or refuse prior standard treatment regimens. At least 1 measurable lesion per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
3. Life expectancy ≥ 3 months.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1.
5. Adequate organ and bone marrow function. Laboratory tests that meet the following criteria within 7 days prior to the first dose of study treatment (without blood transfusion, erythropoietin, recombinant human thrombopoietin or colony stimulating factor therapy, renal replacement therapy, etc., within 28 days prior to the screening examination):

   Routine blood test:

   Absolute neutrophil count (ANC) ≥ 1.5×109/L Platelets count (PLT) ≥ 100×109/L Hemoglobin (Hb) ≥ 90 g/L

   Hepatic function:

   Total bilirubin (TBIL) ≤ 1.5×ULN Aspartate aminotransferase (AST) ≤ 2.5×ULN Alanine aminotransferase (ALT) ≤ 2.5×ULN ALT and AST ≤ 5×ULN and TBIL ≤ 3×ULN for patients with primary liver cancer, liver metastases, or Gilbert 's syndrome.

   Renal function:

   Creatinine clearance ≥ 50 mL/min (calculated according to Cockcroft-Gault formula).

   Coagulation function:

   International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5×ULN
6. Females and males of childbearing potential must agree to use appropriate methods of contraception (hormonal/barrier method or abstinence) during the study and for 3 months after the last dose. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to administration.

Understand and be willing to sign written informed consent and be able to follow the study protocol for treatment, visits, and other study procedures.

Exclusion Criteria:

* 1.Treated with DNA-PK inhibitors. 2.Patients who have received systemic chemotherapy, traditional Chinese medicine for anti-tumor indications or other anti-tumor drugs (including endocrine therapy, molecular targeted therapy, immunotherapy, biological therapy, etc.) within 4 weeks or 5 half-lives (whichever is longer) prior to the first dose of the study drug, or those who need to continue receiving these drugs during the study, with the following three exceptions: Receiving nitrosourea or mitomycin C, which needs more than 6 weeks from the last dose.

Receiving extensive radiotherapy (> 30% of bone marrow radiation), which needs more than 8 weeks from the last radiotherapy.

History of palliative radiotherapy for bone metastases, which needs more than 2 weeks from the last radiotherapy.

3.Major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of the study drug and surgery is scheduled during the study period.

4.Brain metastasis (except asymptomatic, stable for more than 4 weeks prior to the first dose and not requiring steroid therapy for at least 4 weeks prior to the first dose, no imaging findings of marked edema around the tumor lesion), presence of meningeal metastasis or brainstem metastasis, or presence of spinal cord compression.

5.History of other malignancy within the past 5 years, except skin basal cell carcinoma, skin squamous cell carcinoma, cervical carcinoma in situ, or other carcinomas in situ which have undergone curative treatment and have had no recurrence within 5 years after treatment.

6.Toxicities from prior antitumor therapy that have not recovered to CTCAE version 5.0 Grade 1 or less, except CTCAE (V5.0) Grade 2 peripheral neurotoxicity and alopecia of any grade.

7.Serious or uncontrolled diseases as assessed by the investigator, including but not limited to: Severe or uncontrolled diabetes (fasting blood glucose ≥ 10 mmol/L), poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg under standardized antihypertensive regimens), epilepsy, chronic obstructive pulmonary disease, interstitial pneumonia, pulmonary interstitial fibrosis, Parkinson 's disease, active bleeding, uncontrolled infection.

Cognitive dysfunction, history of psychiatric disorders, other uncontrolled concomitant diseases, alcohol dependence, hormone dependence, or drug abuse.

History of immunodeficiency, including HIV antibody positive, other acquired or congenital immunodeficiency disease, or history of organ transplantation.

HBsAg or HBcAb positive, and peripheral blood HBV DNA titer test ≥ 200 IU/mL or ≥ 1000 copies/mL or above the upper limit of normal value at the study site; HCV antibody test positive, and HCV RNA test above the upper limit of normal value at the study site; treponema pallidum-specific antibody positive.

Clinically serious gastrointestinal dysfunction that may compromise drug intake, transport, or absorption. For example, inability to take oral medication, uncontrollable nausea or vomiting, history of massive gastrointestinal resection, history of gastrointestinal ulcer and gastrointestinal bleeding within 6 months prior to the first dose, untreated recurrent diarrhea, untreated stomach disease requiring long-term use of PPI acid suppressants, Crohn 's disease, ulcerative colitis, etc.

Prior thyroid dysfunction or inability to maintain thyroid function within normal limits even with medical therapy.

8.Cardiac dysfunction, including any of the following: Myocardial infarction in past 6 months, heart failure classified as Class II/III/IV according to the New York Heart Association (NYHA) Functional Classification, unstable angina pectoris, and unstable arrhythmia.

Left ventricular ejection fraction LVEF < 50% shown by echocardiography. QT interval corrected using Fridericia 's formula: QTcF > 470 msec (females), QTcF > 450 msec (males).

9.Pregnant (positive pregnancy test prior to dosing) or lactating. 10.History of serious hypersensitivity (e.g., anaphylactic shock) or hypersensitivity to excipients or other ingredients associated with the study drug.

Other factors considered unsuitable for study enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of BY101298 in patients with advanced solid tumors | through study completion (an average of 1.5 years)
  Grade and frequency of adverse events and serious adverse events
To assess the maximum tolerated dose (MTD) | through study completion (an average of 1.5 years)
  Incidence of Dose limiting Toxicities (DLTs)

SECONDARY OUTCOMES:
To assess preliminary antitumor activity of BY101298 in patients with advanced solid tumors | through study completion (an average of 1.5 years)
  ORR
To assess pharmacokinetics (PK) parameters of BY101298 in patients with advanced solid tumors | through study completion (an average of 1.5 years)
  AUC
To assess pharmacokinetics (PK) parameters of BY101298 in patients with advanced solid tumors | through study completion (an average of 1.5 years)
  Cmax
To assess pharmacokinetics (PK) parameters of BY101298 in patients with advanced solid tumors | through study completion (an average of 1.5 years)
  T1/2

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Affiliated to Shandong First Medical University / Shandong Cancer Research Institute / Shandong Cancer Hospital, Jinan, Shandong, China